CLINICAL TRIAL: NCT05777174
Title: An Open Label, Multi-Center, Safety and Pharmacokinetic Bridging Study of MB-102 (Relmapirazin) and the Use of the MediBeacon® Transdermal GFR Measurement System Using the TGFR Reusable Sensor With Disposable Adhesive Ring in Normal and Renal Compromised Subjects for the Evaluation of Kidney Function
Brief Title: Study of MB-102 (Relmapirazin) and the Use of the MediBeacon® Transdermal GFR Measurement System Using the TGFR Reusable Sensor With Disposable Adhesive Ring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 100-201
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Kidney Diseases; Kidney Injury; Kidney Failure
Keywords: Glomerular Filtration Rate; Relmapirazin; Iohexol; Pharmacokinetics; Transdermal fluorescence detection; MB-102
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — relmapirazin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Participants with eGFR ≥ 70 mL/min/1.73 m^2 (Experimental): A TGFR Reusable Sensor with Disposable Adhesive Ring was placed on participants' chests at least 15 minutes prior to dosing on treatment day, and the MediBeacon Transdermal GFR System was initiated to collect background fluorescence. After the collection of background fluorescence, a single dose of MB-102 (130 mg) was administered intravenously to participants with estimated glomerular filtration rate (eGFR) eGFR ≥ 70 mL/min/1.73 m^2. Approximately half of the participants had Fitzpatrick Scale Type I, II or III, and half had Type IV, V and VI skin color type. Blood samples and fluorescent measurements were collected over 12 hours.
  Interventions: Drug: MB-102; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)
- Participants with eGFR < 70 mL/min/1.73 m^2 (Experimental): A TGFR Reusable Sensor with Disposable Adhesive Ring was placed on participants' chests at least 15 minutes prior to dosing on treatment day, and the MediBeacon Transdermal GFR System was initiated to collect background fluorescence. After the collection of background fluorescence, a single dose of MB-102 (130 mg) was administered intravenously to participants with estimated glomerular filtration rate eGFR < 70 mL/min/1.73 m^2. Approximately half of the participants had Fitzpatrick Scale Type I, II or III, and half had Type IV, V and VI skin color type. Blood samples and fluorescent measurements were collected over 24 hours.
  Interventions: Drug: MB-102; Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR)

INTERVENTIONS:
Drug: MB-102 — 18.6 mg/mL in a 7.0 mL volume administered by intravenous injection over 30 - 60 seconds, followed by a 10 mL normal saline flush administered intravenously over 30 - 60 seconds
  Other Names: Relmapirazin
Device: MediBeacon Transdermal Glomerular Filtration Rate Measurement System (TGFR) — On treatment day, participants had the TGFR reusable sensor with disposable adhesive ring placed on their chest, and the MediBeacon® Transdermal GFR Measurement System was initiated to collect background fluorescence. When this was completed, participants received a single dose of MB-102. Fluorescent measurements were collected for 12-24 hours. For those with significant renal compromise, fluorescent measurements were continued until the sensor no longer detected MB-102 in the body.

SUMMARY:
The goal of this clinical trial was to compare transdermal glomerular filtration rate (tGFR) to plasma-derived indexed GFR (nGFR) using MB-102 (relmapirazin) as the fluorescent compound. Adults with kidney function ranging from estimated glomerular filtration rate (eGFR) <120 to >15 mL/min/1.73 m2 and spanning the entire range of human skin colors as defined by the Fitzpatrick Skin Scale (FSS) were included in the study.

The main questions that the study aimed to answer were:

* To establish that the MB-102 transdermal fluorescence assessed GFR using the MediBeacon Transdermal GFR System with the TGFR reusable sensor with disposable adhesive ring was comparable to the measured MB-102 plasma GFR.
* To evaluate the safety and effectiveness of the MediBeacon Transdermal GFR System and the TGFR reusable sensor with disposable adhesive ring for the non-invasive transdermal fluorescence detection of MB-102 in participants

On dosing day, participants had the TGFR reusable sensor with disposable adhesive ring placed on their chest, and the MediBeacon Transdermal GFR System initiated to collect background fluorescence. When this was completed, participants then received a single dose of MB-102. Blood samples were collected and fluorescent measurements were taken over a 12- or 24-hour (or longer) period, depending upon enrollment group. For those with significant renal compromise, fluorescent measurements were continued until the sensor no longer detected MB-102 in the body. Following completion of the treatment period, participants returned to the study center approximately 1 week later for a safety follow-up visit. Researchers compared the results to see if the transdermal GFR measurements were comparable to the measured plasma GFR.

ELIGIBILITY:
Inclusion Criteria:

* Eligible female non-pregnant participants who are either not of child-bearing potential or willing to use adequate contraception during the trial
* Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose
* For women of childbearing potential, the participant should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
* Men will not donate sperm during the study and for 1 month following the last dose of study drug.
* Participants who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
* Adequate venous access sufficient to allow blood sampling per protocol requirements

Exclusion Criteria:

* Participants positive for COVID-19 at the time of dosing
* Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
* Non-steroidal anti-inflammatory (NSAID) use within 3 days of MB-102 dosing
* The participant has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer).
* History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
* History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (intolerance to a drug is not considered a drug allergy).
* Any characteristics which, in the opinion of the investigator, makes the participant a poor candidate for participation in the clinical trial
* Significant scaring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin
* Use of tanning sprays, tanning products etc. on the upper chest within 2 weeks of dosing day
* Use make-up, lotions, Vaseline or other products on the area of the upper chest on the day prior to or the day of dosing
* Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the participant's ability to complete study requirements or may put the participant at increased risk or compromise the interpretability of study results.
* Currently receiving dialysis
* Currently anuric
* Positive serum pregnancy test
* Participants with an eGFR > 120 mL/min/1.73m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research by Design, LLC, Chicago, Illinois
  - Centricity Research, Columbus, Ohio
  - PPD, Austin, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Period: Overall Study
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2
Started | 84 | 65
Completed | 84 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2 | Total
Number analyzed (Participants) | 84 | 65 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.9) | 66.0 (8.62) | 57.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 47 | 32 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 26 | 60
  Not Hispanic or Latino | 50 | 39 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Black or African American | 26 | 31 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 52 | 30 | 82
  Other | 2 | 2 | 4
  Unknown or not reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Transdermal Derived Glomerular Filtration Rate (tGFR) to the Plasma-derived Indexed Glomerular Filtration Rate (nGFR)
Description: The performance measure of P30 is defined as the proportion of transdermal derived GFR values that are within 30% of the measured plasma-derived GFR across all participants. The comparison of transdermal derived glomerular filtration rate (tGFR) with respect to the plasma-derived indexed glomerular filtration rate (nGFR) was calculated with a double-sided 97% confidence interval (CI). The performance goal was 0.85, and success for the study was defined as a lower limit of the 97% CI greater than 0.85.
Time Frame: Up to 24 hours following the study dose
Population: Modified intent-to-measure population (all participants enrolled in the study for whom an average session tGFR or an average snapshot tGFR had been calculated, with no major protocol deviations and no outlier pharmacokinetic parameters)
Measure: Number (97% Confidence Interval); unit: Proportion of tGFR within 30% of nGFR
Units Other Than Participants: tGFR values
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2
Number analyzed (Participants) | 40 | 35
Number analyzed (tGFR values) | 40 | 35
Proportion of tGFR within 30% of nGFR | 0.950 [0.817 to 0.995] | 0.971 [0.836 to 1.00]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Associated With MB-102 Administration
Description: An adverse event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, temporally associated with the use of a medicinal product, whether or not related to the investigational medical device or drug.
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2
Number analyzed (Participants) | 84 | 65
Participants | 1 | 1

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Associated With the MediBeacon Transdermal GFR Measurement System Device
Description: as for outcome 2
Time Frame: From the time of dosing through the follow-up visit, up to 10 days
Population: Safety Population: all participants who enrolled in the study and were dosed with MB-102
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2
Number analyzed (Participants) | 84 | 65
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the time of dosing through the follow-up visit, up to 10 days
Arm/Group | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 | Participants With eGFR < 70 mL/Min/1.73 m^2
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/65
Other Adverse Events (participants affected / at risk) | 2/84 | 5/65
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With eGFR ≥ 70 mL/Min/1.73 m^2 (N=84) | Participants With eGFR < 70 mL/Min/1.73 m^2 (N=65)
INJECTION SITE EXTRAVASATION (General disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MediBeacon requests that no presentation/publication occur until after the first publication of study results or until 1 yr after a study is completed/terminated early, whichever occurs first. Proposed results publication/disclosure must be given to Sponsor for review at least 45 days prior to the date of submission. If a patent application is to be filed, both the Institution and the Sponsor will defer publication or other disclosure for a period of time, not to exceed an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT05777174/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT05777174/SAP_001.pdf